CLINICAL TRIAL: NCT04654000
Title: Efficacy of Rheopheresis as Adjuvant Treatment of Calciphylaxis in Hemodialysis Patients : a Prospective Randomized Controled Single-blind Trial
Brief Title: Rheopheresis as Adjuvant Treatment of Calciphylaxis
Acronym: RHEO-CAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020_05; 2020-A02896-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-12-02; First posted 2020-12-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Disorder; End Stage Renal Disease; Rare Diseases
Keywords: Calciphylaxis; Rheopheresis; Hemodialysis; Chronic kidney disease
MeSH Terms: conditions — Metabolic Diseases; Kidney Failure, Chronic; Rare Diseases; Calciphylaxis; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheopheresis group (Experimental): In addition to the standards of care, the experimental group will carry out the rheopheresis in two stages:
  * Stage 1: induction treatment: 3 apheresis sessions during the first week (w0; i.e. between D1 and D7) and then 2 apheresis sessions each week for 3 weeks (from w1 to w3; i.e. between D8 and D28) ;
  * Step 2: maintenance treatment with 1 apheresis session per week until the 11th week (i.e. between D29 and D84).
  Interventions: Procedure: Rheopheresis procedure
- Sham-apheresis group (Sham Comparator): In addition to the standards of care, the comparator group will carry out Sham-apheresis sessions according to the same scheme as the rheopheresis sessions of the experimental group.
  Interventions: Procedure: Sham-apheresis

INTERVENTIONS:
Procedure: Rheopheresis procedure — rheopheresis is performed using an automated monitor (Plasauto, company HemaT) in a double-filtration cascade. Plasma purify from of high molecular weight proteins
  Arms: Rheopheresis group
Procedure: Sham-apheresis — Sham-apheresis is performed with the same automated monitor (Plasauto, HemaT company). Extracted plasma is not treated through the secondary filter (Rheofilter) and return to the patient.
  Arms: Sham-apheresis group

SUMMARY:
The investigators propose to set up a prospective randomized controlled trial to control the security and assess the efficacy of adjuvant treatment by rheopheresis in necrotizing-ulcered calciphylaxis in the hemodialysis population.

DETAILED DESCRIPTION:
Calciphylaxis, also known as uremic calcifying arteriolopathy (UCA), is a rare disease that causes painful ischemic skin lesions due to microvascular calcification and thrombosis of the dermis and subcutaneous adipose tissue. Patients with end-stage renal disease (ESRD) are the main target for calciphylaxis. Rheopheresis is a therapeutic apheresis to treat microcirculatory disorders. This double filtration plasmapheresis eliminates a defined spectrum of high molecular weight proteins from human plasma including relevant factors for vascular inflammation and thrombose. The investigators propose a prospective randomized controlled trial to compared the efficacy of rheopheresis as adjuvant treatment to the standard of care compared to standard care with Sham-apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Calciphylaxis with at least one ulcerated or necrotizing lesion
* End stage renal disease requiring hemodialysis
* Weight superior to 30kg
* Subject affiliated to or beneficiary of a social security system
* Subject having signed written informed consent

A patient with progressing calciphylaxis to ulcerate or necrosis despite conventional treatment may also be included.

Exclusion Criteria:

* KARNOFSKY Performance Status Scale inferior to 30%
* Life expectancy (independently of calciphylaxis) estimated < 6 months according to a referring physician expert in hemodialysis
* Uncontrolled infection (persistence of fever despite appropriate antibiotic therapy)
* Common variable immunodeficiency
* Albumin allergy
* Contra-indication to stop anti-vitamin K treatment
* Severe cognitive or psychiatric disorders, patients unable to give an informed consent or unwilling to participate in the study
* Pregnancy or breastfeeding and all the other categories of people with special protection according to the French Code de la Santé Publique (CSP): patients under legal supervision, patients hospitalized without contentment, patients admitted in social or sanitary structures for care and not research, and patients in emergency situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete wound healing of the calciphylaxis-mediated ischemic lesions after 12 weeks of rheopheresis treatment (a total of 17 sessions). | at 12 weeks of treatement
  Complete wound healing is defined as the absence of livedoid peri-lesional inflammation with presence of granulation tissue (stage 3 healing process) and/or epithelization (stage 4) over the entire ulcer surface of calciphylactic lesions. The healing of the lesions will be illustrated with a photographic support. And the pictures will be examined a second time in a centralized and blind way by two referring dermatologists.
  In case of multiple calciphylaxis skin lesions, monitoring and evaluation will be done on the largest lesion at the time of patient's inclusion.

SECONDARY OUTCOMES:
Percentage of patient with partial wound healing of the calciphylaxis mediated lesions after rheopheresis treatment. | At 4 weeks and 12 weeks of rheopheresis treatment.
  The partial healing is defined by a partial reepithelialization (validated if 3 of following 4 criteria are present: 1-absence of necrosis; 2- granulation; 3 less inflammatory bordering 4- 20% decrease of the lesion size). The evolution of the size of the lesions and the partial healing of the wound will be illustrated by a photographic support.
Occurrence of new ulcerated calciphylaxis lesions | At 4 weeks and 12 weeks of rheopheresis treatment.
  Occurrence of new ulcerated calciphyalxis lesions frome Baseline to 4 and 12 weeks of treatment.
Evolution of the self-reporting pain using Numeric Rating Scale (NRS) | from baseline (V0) to 12 weeks of rheopheresis (V2)
  The Numeric Rating Scale (NRS) describes the pain intensity at 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme
Evolution of the level of antalgic consumed according to World Health Organisation (WHO) classification | from baseline (V0) to 12 weeks of rheopheresis (V2)
  The level of consumed antalgic is defined according to the World Health Organization (WHO) classification
  * Level I analgesics = peripheral analgesics or not morphine have the lowest analgesic power
  * Level II analgesics = weak morphine.
  * Level III analgesics = strong morphine agonists and antagonists.
Number of days without antibiotics | during the 12 weeks of rheopheresis treatment
  Number of days the patient receives antibiotics, regardless of the route of administration, whether the patient is treated on an outpatient or inpatient basis.
Quality of life by the Wound quality of life score (Wound-Qol) | form baseline (V0) and at 12 weeks
  The Wound-QoL measures the disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which are always assessed in retrospect to the preceding seven days.
Number of days discharged from hospital | during the 12 weeks of rheopheresis treatment
  Number of days the patient is treated on an outpatient basis.
Overall survival | at 12 weeks and 12 months after first rheopheresis.
  Survival of patients, whether or not calciphylaxis is cured.
Change in inflammatory proteins | from baseline to 12 weeks-rheopheresis treatment
  Change in the plasmatic rates of C-reactive protein (CRP) and fibrinogen.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Lionet, MD, Principal Investigator — University Hospital, Lille
Locations (29):
- France (29):
  - CHU d'Angers, Angers
  - CHU d'Arras, Arras
  - CHU d'Auxerre, Auxerre
  - CHU de Besançon, Hôpital Jean Minjoz, Besançon
  - CH de Béthune, Béthune
  - CH de Boulogne sur Mer, Boulogne-sur-Mer
  - CHU de Bordeaux, Bourdeaux
  - CHRU de Brest, Brest
  - CHU de Caen, Caen
  - Hôpital Nord Michallon, CHU de Grenoble, Grenoble
  - Centre ECHO Laval, Laval
  - Centre ECHO Le Mans, Le Mans
  - Hôpital Privé La Louvière, Lille
  - Hop Claude Huriez Chu Lille, Lille
  - CHR de Limoges, Limoges
  - Hôpital Lyon Sud, Lyon
  - Hôpital Saint Joseph Saint Luc, Lyon
  - Institut Phocéen de Néphrologie - Clinique Bouchard, Marseille
  - Hôpital de la Conception, AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CH de Niort, Niort
  - CHU de Reims, Reims
  - CHU de Toulouse, Toulouse
  - Clinique Saint Exupéry, Toulouse
  - CH de Valenciennes, Valenciennes
  - CHRU de Nancy Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - CH de Vichy, Vichy